CLINICAL TRIAL: NCT02701985
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Phase 2A Study to Assess the Efficacy of RO5459072 in Patients With Primary Sjogren's Syndrome
Brief Title: A Study to Assess the Efficacy of RO5459072 in Participants With Primary Sjogren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP30037; 2015-004476-30 (EudraCT Number)
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — petesicatib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Matching-placebo capsules will be administered orally, 2 times a day, for up to 12 weeks.
  Interventions: Drug: Placebo
- RO5459072 (Experimental): RO5459072 at a dose of 100 milligrams (as capsules) will be administered orally, 2 times a day, for up to 12 weeks.
  Interventions: Drug: RO5459072

INTERVENTIONS:
Drug: Placebo — Matching-placebo capsules will be administered orally, 2 times a day with food.
  Arms: Placebo
Drug: RO5459072 — RO5459072 at a dose of 100 milligrams (as capsules) will be administered orally, 2 times a day with food.
  Arms: RO5459072

SUMMARY:
This is a randomized, double-blind, placebo-controlled, two-treatment arm, parallel-group study designed to evaluate the effects of RO5459072 treatment on disease activity and symptoms of Sjogren's syndrome in adult participants with moderate to severe primary Sjogren's syndrome. The total duration of the study for each participant will be approximately 18 weeks (including screening).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of primary Sjogren's syndrome according to the revised American-European Consensus Group (AECG) criteria
* ESSDAI score greater than or equal to (>/=) 5
* ESSPRI score >/=5
* Elevated serum titers of anti-Sjogren's-syndrome-related antigen A (anti-SSA) and/or anti-Sjogren's-syndrome-related antigen B (anti-SSB) antibodies at screening
* Negative pregnancy test at screening and baseline (for women only)
* Willing to comply with the study procedures and restrictions, including measures to prevent pregnancy and restrictions on sperm donation

Exclusion Criteria:

* A diagnosis of secondary Sjogren's syndrome according to the revised AECG criteria
* Severe complications of Sjogren's syndrome
* Systemic immunosuppressant therapy, cyclophosphamide, or B-cell depleting therapy within 6 months prior to the screening visit
* Corticosteroid therapy exceeding 7.5 mg prednisone equivalents per day
* A positive test result for hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV), or tuberculosis, or any other active viral, fungal, yeast or bacterial infection at screening
* A history suggesting reduced immune function or any other conditions predisposing participants to serious infection
* A history of lymphoma, myeloma or monoclonal gammopathy of unknown significance (MGUS), or any other malignancies within the past 5 years
* A diagnosis of fibromyalgia or significant depression
* Having any concomitant disease or condition that could interfere with the conduct of the study, or that would pose an unacceptable risk to the individual
* Participation in an investigational drug or device study within 3 months prior to screening
* Inability to comply with the study protocol for any other reason
* Women who are lactating, breastfeeding or planning to nurse
* Using other prohibited medication (moderate or potent inhibitors of CYP3A4; strong inducers of CYP3A4; strong inhibitors of the transporter P-glycoprotein [P-gp]; sensitive substrates of CYP3A4 with a narrow therapeutic index)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- United States (12):
  - Wallace Rheumatic Study Center, Beverly Hills, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - John Hopkins Bayview Medical Center, Baltimore, Maryland
  - University Of Michigan, Ann Arbor, Michigan
  - Winthrop University Hospital, Mineola, New York
  - Shanahan Rheumatology & Immunology, PLLC, Raleigh, North Carolina
  - MetroHealth System, Cleveland, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Ramesh Gupta - PP, Memphis, Tennessee
- France (4):
  - Hopital Avicenne, Paris, Bobigny
  - C.H.U. Ambroise Pare (AP-HP), Boulogne-Billancourt
  - Hopital La Cavale Blanche; Rhumatologie, Brest
  - Hopital Lapeyronie; Immunologie Rhumatologie, Montpellier
- Charité Research Organisation GmbH, Berlin, Germany
- Poland (4):
  - Szpital Uniwersytecki; nr 2 im. Dr J. Biziela; Klinika Reumatologii i Ukladowych Chorob, Bydgoszcz
  - MedPolonia, Poznan
  - Niepubliczny Opieki Zdrowotnej; Reumatika - Ctr Reum., Warsaw
  - Centrum Medyczne AMED, Warsaw
- Portugal (4):
  - Instituto Portugues de Reumatologia, Lisbon
  - Centro Hospitalar de Lisboa Norte, EPE - Hospital Santa Maria, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - Centro Hospitalar de Sao Joao,E.P.E., Porto
- United Kingdom (6):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Barts and the London NHS Trust, London
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Sheffield Teaching Hospitals NHS Foundation Trust; Royal Hallamshire Hospital, Sheffield
  - Great Western Hospitals NHS Foundation Trust., Wiltshire

REFERENCES:
- [Derived] Bentley D, Fisher BA, Barone F, Kolb FA, Attley G. A randomized, double-blind, placebo-controlled, parallel group study on the effects of a cathepsin S inhibitor in primary Sjogren's syndrome. Rheumatology (Oxford). 2023 Nov 2;62(11):3644-3653. doi: 10.1093/rheumatology/kead092. PMID 36864622

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 75 patients were randomized in a 1:1 ratio to RO5459072 or placebo (38 patients in the RO5459072 treatment group and 37 patients in the placebo group).
Groups:
- Placebo: Matching-placebo capsules was administered orally, 2 times a day, for up to 12 weeks.
- RO5459072: RO5459072 at a dose of 100 milligrams (as capsules) was administered orally, 2 times a day, for up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo | RO5459072
Started | 37 | 38
Completed | 34 | 32
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | RO5459072 | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.8) | 52.1 (13.2) | 52.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 1 | 6 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 35 | 38 | 73
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 33 | 35 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Clinically Relevant Decrease in European League Against Rheumatism (EULAR) Sjogren's Syndrome Disease Activity Index (ESSDAI) Score
Description: Percentage of participants with a clinically relevant decrease in European League Against Rheumatism (EULAR) Sjogren's Syndrome Disease Activity Index (ESSDAI) Score is defined as participants with absolute decrease of ≥ 3-points in ESSDAI score. ESSDAI is physician-assessed disease activity index developed by EULAR consortium consisting of 44 items in 12 organ-specific 'domains' (constitutional,lymphadenopathy, articular,muscular,cutaneous,glandular,pulmonary,renal,peripheral nervous system,central nervous system,hematological,biological). Each domain is assessed for activity level (i.e., no, low, moderate, high) and assigned a numerical score based on pre-determined weighting of each individual domain. Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 (best) to 123 (worst activity). A score ≥ 5 is considered moderate or severe disease activity and a clinically relevant change in ESSDAI score is defined as absolute decrease of ≥ 3-points.
Time Frame: 12 weeks
Population: Modified intent-to-treat (mITT) population was defined as all randomized participants, who received any study medication and had evaluable measurement of the parameter of interest at baseline and at least one post-baseline visit.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
Percentage of Participants | 37.8 [20.86 to 54.86] | 42.1 [25.09 to 59.12]
Statistical Analysis 1: Comparison: Placebo vs RO5459072; The proportion of patients who have ≥ 3 point reduction from baseline in ESSDAI score after 12 weeks of treatment was compared between the two treatment arms using a Pearson Chi-square test (two sided p-values, alpha 0.05). The difference in proportions and corresponding 95% confidence interval (CI) are provided. Patients with missing data at Week 12 will be treated as non-responders in the analysis; Test type: Other; p = 0.7955, Chi-square with Schouten Correction; Difference in Response Rates = 4.27, 95% CI 2-sided [-20.55 to 29.08]

2. Secondary Outcome: Percentage of Participants With a Clinically Relevant Decrease in EULAR Sjogren's Syndrome Patient-Reported Index (ESSPRI) Score
Description: The efficacy of RO5459072 in patients with primary Sjogren's Syndrome Disease is evaluated in terms of the percentage of participants with a clinically relevant decrease in EULAR Sjogren's Syndrome Patient-Reported Index (ESSPRI) Score, where a clinically relevant decrease in ESSPRI score is defined as a decrease of ≥ 1 point. The ESSPRI is a patient-reported, subjective symptom index for primary Sjögren's syndrome developed by the EULAR consortium. It consists of 3 questions covering cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain (articular and/or muscular). Each domain scored on scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable), and overall score is calculated as the mean of 3 individual domains where all domains carry same weight.
Time Frame: 12 weeks
Population: mITT population was defined as all randomized participants, who received any study medication and had evaluable measument of the parameter of interest at baseline and at least one post-baseline visit.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
Percentage of Participants | 56.8 [39.44 to 74.07] | 57.9 [40.88 to 74.91]
Statistical Analysis 1: Comparison: Placebo vs RO5459072; The proportion of patients who have ≥ 1 point reduction from baseline in ESSPRI score after 12 weeks of treatment was compared between the two treatment arms using a Pearson Chi-square test (two sided p-values, alpha 0.05). The difference in proportions and corresponding 95% CI are provided. Patients with missing data at Week 12 will be treated as non-responders in the analysis; Test type: Other; p = 0.9877, Chi-square with Schouten Correction; Difference in Response Rates = 1.14, 95% CI 2-sided [-23.92 to 26.19]

3. Secondary Outcome: Change From Baseline in ESSDAI Score at Week 12
Description: Change from baseline in European League Against Rheumatism (EULAR) Sjogren's Syndrome Disease Activity Index (ESSDAI) Score is defined as the change in score between baseline (Week -1) and Week 12. The ESSDAI is a physician-assessed disease activity index for primary Sjögren's syndrome developed by the EULAR consortium. It consists of 44 items in 12 organ-specific 'domains' contributing to disease activity (constitutional, lymphadenopathy, articular, muscular, cutaneous, glandular, pulmonary, renal, peripheral nervous system, central nervous system, hematological, biological). Each domain is assessed for activity level (i.e., no, low, moderate, high) and assigned a numerical score based on pre-determined weighting of each individual domain. An overall score is then calculated as the sum of all individual weighted domain scores. Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 (best) to 123 (worst activity).
Time Frame: Baseline (Week -1), Week 12
Population: mITT population was defined as all randomized participants, who received any study medication and had evaluable measurement of the parameter of interest at baseline and at least one post-baseline visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
scores on a scale
  Baseline in ESSDAI Score | 11.27 (5.71) | 11.79 (4.69)
  Change From Baseline in ESSDAI Score at Week 12 | -3.06 (3.96) | -3.25 (4.09)
Statistical Analysis 1: Comparison: Placebo vs RO5459072; A Mixed Model for Repeated Measures (MMRM) approach incorporating all observed data up to 12 weeks of treatment was used. The MMRM included the absolute change from baseline as the dependent variable; Test type: Superiority; p = 0.8905, Mixed Model for Repeated Measures; Difference in Adjusted Means = -0.13, 95% CI 2-sided [-2.04 to 1.78]

4. Secondary Outcome: Change From Baseline in ESSPRI Score at Week 12
Description: Change from baseline in EULAR Sjogren's Syndrome Patient-Reported Index (ESSPRI) Score is defined as the change in score between baseline (Week -1) and Week 12. The ESSPRI is a patient-reported, subjective symptom index for primary Sjögren's syndrome developed by the EULAR consortium. It consists of three questions covering the cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain (articular and/or muscular). Each domain scored on scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable), and an overall score is calculated as the mean of the three individual domains where all domains carry the same weight.
Time Frame: Baseline (Week -1), Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
Score on a scale
  Baseline in ESSPRI Score | 7.34 (1.19) | 6.98 (0.98)
  Change From Baseline in ESSPRI Score at Week 12: number analyzed (Participants) | 34 | 32
  Change From Baseline in ESSPRI Score at Week 12 | -1.35 (1.67) | -1.51 (1.79)
Statistical Analysis 1: Comparison: Placebo vs RO5459072; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.6077, Mixed Model of Repeated Measures; Difference in Adjusted Means = -0.22, 95% CI 2-sided [-1.08 to 0.64]

5. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36) Mental Score at Week 12
Description: Change from baseline in Short Form-36 Health Survey (SF-36) Mental score is defined as the change in score between baseline (Week -1) and Week 12. The SF-36 was used to assess health-related quality of life at baseline and at on-treatment visits. The SF-36 consisted of 36 questions covering 8 domains (general health, physical functioning, role-functioning physical, bodily pain, social functioning, role-functioning emotional, mental health, and vitality), with each domain scoring on a scale 0-100 (a score of 0 = maximum disability and a score of 100 = no disability). Reported here is the mental health domain score.
Time Frame: Baseline (Week -1), Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
Score on a scale
  Baseline: number analyzed (Participants) | 35 | 37
  Baseline | 42.09 (11.18) | 40.52 (9.27)
  Change from Baseline at Week 12: number analyzed (Participants) | 32 | 31
  Change from Baseline at Week 12 | 4.52 (7.15) | 3.02 (9.04)
Statistical Analysis 1: Comparison: Placebo vs RO5459072; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.2846, Mixed Model of Repeated Measures; Difference in Adjusted Means = -2.06, 95% CI [-5.87 to 1.75]

6. Secondary Outcome: Change From Baseline in SF-36 Physical Score at Week 12
Description: Change from baseline in Short Form-36 Health Survey (SF-36) Physical Score is defined as the change in score between baseline (Week -1) and Week 12. The SF-36 was used to assess health-related quality of life at baseline and at on-treatment visits. The SF-36 consisted of 36 questions covering 8 domains (general health, physical functioning, role-functioning physical, bodily pain, social functioning, role-functioning emotional, mental health, and vitality), with each domain scoring on a scale 0-100. (a score of 0 = maximum disability and a score of 100 = no disability)
Time Frame: Baseline (Week -1), Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
Score on a scale
  Baseline in SF-36 Physical Score: number analyzed (Participants) | 35 | 37
  Baseline in SF-36 Physical Score | 40.86 (6.82) | 40.71 (6.94)
  Change From Baseline at Week 12: number analyzed (Participants) | 32 | 31
  Change From Baseline at Week 12 | 2.46 (6.09) | 3.01 (5.10)
Statistical Analysis 1: Comparison: Placebo vs RO5459072; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.8134, Mixed Model of Repeated Measures; Difference in Adjusted Means = -0.33, 95% CI [-2.43 to 3.08]

7. Secondary Outcome: Change From Baseline in ESSPRI Dryness Component Score at Week 12
Description: Change from baseline in EULAR Sjogren's Syndrome Patient-Reported Index (ESSPRI) dryness component score is defined as the change in score between baseline (Week -1) and Week 12. The Dryness Component score ranged from 0-10 (0 =no symptom at all and 10 = worst symptom imaginable).
Time Frame: Baseline (Week -1), Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
Score on a scale
  Baseline | 7.54 (1.57) | 7.45 (1.25)
  Change From Baseline at Week 12: number analyzed (Participants) | 34 | 31
  Change From Baseline at Week 12 | -1.15 (1.56) | -1.77 (2.29)

8. Secondary Outcome: Change From Baseline in ESSPRI Fatigue Component Score at Week 12
Description: Change from baseline in EULAR Sjogren's Syndrome Patient-Reported Index (ESSPRI) fatigue component score is defined as the change in score between baseline (Week -1) and Week 12. The ESSPRI score consists of three questions covering the cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain (articular and/or muscular). Each domain scored on scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable).
Time Frame: Baseline (Week -1), Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
Score on a scale
  Baseline | 7.22 (1.81) | 7.24 (1.84)
  Change From Baseline at Week 12: number analyzed (Participants) | 34 | 31
  Change From Baseline at Week 12 | -1.29 (2.24) | -1.94 (2.16)

9. Secondary Outcome: Change From Baseline in EULAR Sjogren's Syndrome Patient-Reported Index (ESSPRI) Pain Component Score at Week 12
Description: Change from baseline in EULAR Sjogren's Syndrome Patient-Reported Index (ESSPRI) pain component score is defined as the change in score between baseline (Week -1) and Week 12. The ESSPRI score consists of three questions covering the cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain (articular and/or muscular). Each domain scored on scale of 0-10 (Each domain scored on scale of 0-10 (0 = no symptom at all and 10 = worst symptom imaginable).
Time Frame: Baseline (Week -1), Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
Score on a scale
  Baseline | 7.27 (1.71) | 6.26 (2.05)
  Change From Baseline at Week 12: number analyzed (Participants) | 34 | 31
  Change From Baseline at Week 12 | -1.62 (2.70) | -0.97 (2.56)

10. Secondary Outcome: Change From Baseline in Tear Flow Rate at Weeks 2, 6, and 12
Description: Un-stimulated tear production rate was measured from both eyes (without the use of analgesics/ anesthetic drops) at baseline and at on-treatment visits using the Schirmer method. A thin strip of filter paper (Schirmer strip, e.g., 35 x 5 mm) was placed at the junction of the lateral and middle thirds of the lower eyelid of each eye. The maximum length of wetting along the strip at the end of the test period was measured.
Time Frame: Baseline, Week 2, Week 6, and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/5 min
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
mm/5 min
  Baseline in Tear Flow Rate | 7.53 (9.66) | 7.84 (10.15)
  Change from Baseline at Week 2: number analyzed (Participants) | 37 | 34
  Change from Baseline at Week 2 | -0.54 (5.02) | -0.81 (5.06)
  Change from Baseline at Week 6: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 6 | -1.39 (6.32) | -0.95 (7.95)
  Change from Baseline at Week 12: number analyzed (Participants) | 34 | 30
  Change from Baseline at Week 12 | -2.38 (6.47) | -1.65 (7.71)
Statistical Analysis 1: Comparison: Placebo vs RO5459072; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4266, Mixed Model of Repeated Measures; Median Difference (Final Values) = 0.87, 95% CI [-1.30 to 3.03]

11. Secondary Outcome: Change From Baseline in Mechanically Stimulated Salivary Flow Rate at Weeks 2, 6, and 12
Description: Change from baseline in mechanically stimulated salivary flow rate is defined as the change in flow (mL/min) between baseline (Week -1) and Week 2, Week 6 and Week 12. Using a mechanical stimulation method of a piece of neutral wax, paraffin, silicone, unflavored chewing gum, or similar chewable, unflavored, nonabsorbent material, patients were instructed to chew for a period of 5 minutes. The stimulated salivary flow rate was calculated assuming a specific gravity of 1 (i.e., 1 mL saliva = 1 g) and expressed in mL per minute.
Time Frame: Baseline, Week 2, Week 6, and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
mL/min
  Baseline | 0.45 (0.29) | 0.55 (0.58)
  Change from Baseline at Week 2: number analyzed (Participants) | 37 | 34
  Change from Baseline at Week 2 | 0.10 (0.33) | -0.01 (0.33)
  Change from Baseline at Week 6: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 6 | 0.10 (0.31) | 0.11 (0.47)
  Change from Baseline at Week 12: number analyzed (Participants) | 34 | 31
  Change from Baseline at Week 12 | 0.12 (0.30) | 0.24 (0.75)
Statistical Analysis 1: Comparison: Placebo vs RO5459072; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.6429, Mixed Model of Repeated Measures; Mean Difference (Final Values) = 0.06, 95% CI [-0.21 to 0.34]

12. Secondary Outcome: Change From Baseline in Anti-Sjögren's-Syndrome-Related Antigen A at Weeks 6, and 12
Description: Anti-Sjögren's-syndrome-related antigen A is a type of antibody found in the auto-antibody titers.
Time Frame: Baseline, Week 6, and Week 12
Population: The safety population included all participants, who received at least one dose of the study medication. Participants were grouped according to the treatment actually received.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
U/mL
  Baseline | 214.52 (58.06) | 217.78 (53.96)
  Change from Baseline at Week 6: number analyzed (Participants) | 35 | 33
  Change from Baseline at Week 6 | -4.82 (16.05) | -1.47 (13.90)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 31
  Change from Baseline at Week 12 | -2.57 (18.97) | -5.20 (11.65)

13. Secondary Outcome: Change From Baseline in Anti-Sjögren's-Syndrome-Related Antigen B at Weeks 6, and 12
Description: Anti-Sjögren's-syndrome-related antigen B is a type of antibody found in the auto-antibody titers.
Time Frame: Baseline, Week 6, and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
U/mL
  Baseline | 101.66 (130.48) | 76.94 (120.76)
  Change from Baseline at Week 6: number analyzed (Participants) | 35 | 33
  Change from Baseline at Week 6 | 1.94 (15.20) | -2.55 (13.09)
  Change from Baseline at Week 12: number analyzed (Participants) | 33 | 31
  Change from Baseline at Week 12 | 1.35 (13.52) | -4.47 (12.32)

14. Secondary Outcome: Change From Baseline in Rheumatoid Factor at Weeks 6, and 12
Description: Rheumatoid factor is a type of auto-antibody found in the auto-antibody titers.
Time Frame: Baseline, Week 6, and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kU/L
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
kU/L
  Baseline in Rheumatoid Factor | 43.00 (48.51) | 117.84 (336.82)
  Change from Baseline at Week 6: number analyzed (Participants) | 36 | 33
  Change from Baseline at Week 6 | -1.50 (10.74) | -28.03 (70.04)
  Change from Baseline at Week 12: number analyzed (Participants) | 34 | 31
  Change from Baseline at Week 12 | -0.68 (9.97) | -57.77 (173.75)

15. Secondary Outcome: Change From Baseline in Total Immunoglobulin G (IgG) at Weeks 6, and 12
Description: Total IgG is a type of auto-antibody found in the auto-antibody titers.
Time Frame: Baseline, Week 6, and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
g/L
  Baseline in Total IgG | 15.74 (6.77) | 13.59 (4.92)
  Change from Baseline at Week 6: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 6 | 0.11 (1.51) | -0.30 (1.21)
  Change from Baseline at Week 12: number analyzed (Participants) | 34 | 31
  Change from Baseline at Week 12 | 0.48 (1.78) | -0.50 (1.13)

16. Secondary Outcome: Change From Baseline in Total Immunoglobulin M (IgM) at Weeks 6, and 12
Description: Total IgM is a type of auto-antibody found in the auto-antibody titers.
Time Frame: Baseline, Week 6, and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
g/L
  Baseline in Total IgM | 1.24 (0.82) | 1.26 (0.75)
  Change from Baseline at Week 6: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 6 | 0.03 (0.20) | -0.10 (0.17)
  Change from Baseline at Week 12: number analyzed (Participants) | 34 | 30
  Change from Baseline at Week 12 | 0.06 (0.25) | -0.17 (0.20)

17. Secondary Outcome: Minimum Concentration (Cmin) of RO5459072
Description: Minimum observed plasma concentration (mass/volume)
Time Frame: Week 2, Week 6, and Week 12
Population: as for outcome 12
Measure: Median (90% Confidence Interval); unit: ng/mL
Arm/Group | RO5459072
Number analyzed (Participants) | 38
ng/mL | 1340 [2.68 to 2900]

18. Secondary Outcome: Maximum Concentration (Cmax) of RO5459072
Description: Maximum observed plasma concentration (mass/volume)
Time Frame: Week 2, Week 6, and Week 12
Population: as for outcome 12
Measure: Median (90% Confidence Interval); unit: ng/mL
Arm/Group | RO5459072
Number analyzed (Participants) | 38
ng/mL | 2350 [1140 to 3610]

19. Secondary Outcome: Average Concentration (Caverage) of RO5459072
Description: Average observed plasma concentration (mass/volume)
Time Frame: Week 2, Week 6, and Week 12
Population: as for outcome 12
Measure: Median (90% Confidence Interval); unit: ng/mL
Arm/Group | RO5459072
Number analyzed (Participants) | 38
ng/mL | 1740 [816 to 3187]

20. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to Week 14
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | RO5459072
Number analyzed (Participants) | 37 | 38
Percentage of participants | 78.4 | 76.3

ADVERSE EVENTS:
Time Frame: The total duration of the study for each patient was (up to) 19 weeks.
Description: The safety population is defined as all patients who received at least one dose of the study medication.
Arm/Group | Placebo | RO5459072
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 2/37 | 1/38
Other Adverse Events (participants affected / at risk) | 19/37 | 25/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | RO5459072 (N=38)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | RO5459072 (N=38)
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 5
Fatigue (General disorders) | 1 | 2
Pyrexia (General disorders) | 2 | 0
Bronchitis (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 3 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 5
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 | 6
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 4 | 5
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT02701985/Prot_SAP_000.pdf